CLINICAL TRIAL: NCT04530838
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, THIRD PARTY UNBLIND TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN HEALTHY JAPANESE INFANTS
Brief Title: 20-valent Pneumococcal Conjugate Vaccine Safety and Immunogenicity Study in Healthy Japanese Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B7471016; 2022-001146-38 (EudraCT Number)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 20-valent pneumococcal conjugate vaccine (subcutaneous) (Experimental): 20-valent pneumococcal conjugate vaccine administered by subcutaneous injection (SC)
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine
- 13-valent pneumococcal conjugate vaccine (subcutaneous) (Active Comparator): 13-valent pneumococcal conjugate vaccine administered by subcutaneous injection (SC)
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine
- 20-valent pneumococcal conjugate vaccine (intramuscular) (Experimental): 20-valent pneumococcal conjugate vaccine administered by intramuscular injection (IM)
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 20-valent pneumococcal conjugate vaccine — 20-valent pneumococcal conjugate vaccine
  Arms: 20-valent pneumococcal conjugate vaccine (intramuscular); 20-valent pneumococcal conjugate vaccine (subcutaneous)
Biological: 13-valent pneumococcal conjugate vaccine — 13-valent pneumococcal conjugate vaccine
  Arms: 13-valent pneumococcal conjugate vaccine (subcutaneous)

SUMMARY:
20-valent Pneumococcal Conjugate Vaccine Safety and Immunogenicity Study in Healthy Japanese Infants

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or female infants ≥2 months to ≤6 months at the time of consent.
* Healthy infants determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study.

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis)
* Major known congenital malformation or serious chronic disorder.
* History of microbiologically proven invasive disease caused by S pneumoniae.
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 668 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- Japan (38):
  - NHO Nagoya Medical Center, Nagoya, Aichi-ken
  - TOYOTA Memorial Hospital, Toyota-shi, Aichi-ken
  - Tsubaki Children's Clinic, Chiba, Chiba
  - Sunrise Children's Clinic, Funabashi, Chiba
  - medical corporation Shigyo-no-kai Sotobo Children's Clinic, Isumi, Chiba
  - Sou Clinic, Yotsukaido-shi, Chiba
  - NHO Shimoshizu National Hospital, Yotsukaido-shi, Chiba
  - Fukui Aiiku Hospital, Fukui-shi, Fukui
  - Fukazawa Clinic, Fukuoka, Fukuoka
  - Shindo children's clinic, Fukuoka, Fukuoka
  - Shimomura Pediatrics Clinic, Fukuoka, Fukuoka
  - Inamitsu Children's Clinic, Fukuoka, Fukuoka
  - Iizuka Hospital, Iizuka, Fukuoka
  - Yokoyama Children'S Clinic, Kasuga, Fukuoka
  - Yajima Children's Clinic, Gifu, Gifu
  - Azuma kodomo katei clinic, Ebetsu Shi, Hokkaido
  - Nakata pediatric clinic, Sapporo, Hokkaido
  - Nishi Sapporo Pediatrics, Sapporo, Hokkaido
  - Yoshimura Child Clinic, Akashi, Hyōgo
  - Morino Kodomo Clinic, Kawasaki-shi, Kanagawa
  - Sakuranbo Kodomo Clinic, Kumamoto, Kumamoto
  - MIURA Children's Clinic, Kumamoto, Kumamoto
  - Matsuda Pediatric Clinic, Kuwana, Mie-ken
  - Arakawa Family Clinic, Nagano, Nagano
  - NHO Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - Aizenbashi Hospital, Osaka, Osaka
  - NHO Ureshino Medical center, Ureshino-shi, Saga-ken
  - Hanyu General Hospital, Hanyu-shi, Saitama
  - Enomoto Clinic, Kumagaya-shi, Saitama
  - Saiseikai Shiga Hospital, Ritto-Shi, Shiga
  - Sakiyama Pediatric Clinic, Fuchū, Tokyo
  - Saitoh-Clinic, Nishi-Tokyo-shi, Tokyo
  - Inami Pediatrics, Setagaya-ku, Tokyo
  - Sasamoto Children's Clinic, Setagaya-ku, Tokyo
  - Futaba Clinic, Shinjuku-ku, Tokyo
  - Tamura Clinic, Suginami-ku, Tokyo
  - Childrens clinic of Kose, Kofu, Yamanashi
  - Takei Clinic, Tsuru-shi, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Ishihara Y, Fukazawa M, Enomoto S, de Solom R, Yamaji M, Kline M, Aizawa M, Peng Y, Kogawara O, Giardina PC, Tamimi N, Gruber WC, Watson W. A phase 3 randomized study to evaluate safety and immunogenicity of 20-valent pneumococcal conjugate vaccine in healthy Japanese infants. Int J Infect Dis. 2024 Apr;141:106942. doi: 10.1016/j.ijid.2024.01.009. Epub 2024 Jan 17. PMID 38242195
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471016

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 668 participants were enrolled and randomized in the study. One participant did not receive any study vaccine. One participant receive vaccination through route which was not as per randomization. Hence, data of these participants were excluded from analysis.
Groups:
- 20vPnC (SC): Participants received 4 doses of 0.5 milliliter (mL) 20-valent Pneumococcal Conjugate Vaccine (20vPnC) subcutaneously (SC) into the anterolateral thigh. The time interval between Dose 1, 2 and 3 was 4 to 8 weeks from the previous vaccination. Participants completed Dose 1, 2 and 3 by 12 months of age. Dose 4 was administered at least after 60 days of Dose 3.
- 13vPnC (SC): Participants received 4 doses of 0.5 mL 13-valent Pneumococcal Conjugate Vaccine (13vPnC) SC into the anterolateral thigh. The time interval between Dose 1, 2 and 3 was 4 to 8 weeks from the previous vaccination. Participants completed Dose 1, 2 and 3 by 12 months of age. Dose 4 was administered at least after 60 days of Dose 3.
- 20vPnC (IM): Participants received 4 doses of 0.5 mL 20vPnC intramuscularly (IM) into the anterolateral thigh muscle. The time interval between Dose 1, 2 and 3 was 4 to 8 weeks from the previous vaccination. Participants completed Dose 1, 2 and 3 by 12 months of age. Dose 4 was administered at least after 60 days of Dose 3.
Period: Overall Study
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Started | 225 | 224 | 217
Completed | 217 | 220 | 211
Not Completed | 8 | 4 | 6
Not completed — Other | 2 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — No longer meets eligibility criteria | 1 | 0 | 2
Not completed — Withdrawal by parent/guardian | 5 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all the participants who received at least 1 dose of the investigational product (IP) with safety follow up after any vaccination.
Groups:
- 20vPnC (SC): Participants received 4 doses of 0.5 mL 20vPnC SC into the anterolateral thigh. The time interval between Dose 1, 2 and 3 was 4 to 8 weeks from the previous vaccination. Participants completed Dose 1, 2 and 3 by 12 months of age. Dose 4 was administered at least after 60 days of Dose 3.
- 13vPnC (SC): Participants received 4 doses of 0.5 mL 13vPnC SC into the anterolateral thigh. The time interval between Dose 1, 2 and 3 was 4 to 8 weeks from the previous vaccination. Participants completed Dose 1, 2 and 3 by 12 months of age. Dose 4 was administered at least after 60 days of Dose 3.
- 20vPnC (IM): Participants received 4 doses of 0.5 mL 20vPnC IM into the anterolateral thigh muscle. The time interval between Dose 1, 2 and 3 was 4 to 8 weeks from the previous vaccination. Participants completed Dose 1, 2 and 3 by 12 months of age. Dose 4 was administered at least after 60 days of Dose 3.
- Total: Total of all reporting groups
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM) | Total
Number analyzed (Participants) | 225 | 224 | 217 | 666
Age, Continuous [Mean (Standard Deviation); unit: Months] | 2.4 (0.33) | 2.4 (0.40) | 2.4 (0.42) | 2.4 (0.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 114 | 106 | 337
  Male | 108 | 110 | 111 | 329
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 225 | 224 | 217 | 666
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 225 | 224 | 217 | 666
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions (LR) Within 7 Days After Dose 1
Description: Local reactions included pain at injection site, redness and swelling were measured and recorded in measuring device (caliper) units. 1 measuring device unit =0.5 centimeter (cm). Pain at injection site was graded as mild: hurts if gently touched; moderate: hurts if gently touched with crying; severe: limited limb movement. Redness and swelling were graded as mild: >0 to 2.0 cm; moderate >2.0 to 7.0 cm; and severe: >7.0 cm.
Time Frame: Within 7 Days after Dose 1
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after Dose 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 225 | 224 | 217
Percentage of participants
  Redness: Mild | 58.2 (51.5) [51.5 to 64.7] | 51.3 (44.6) [44.6 to 58.1] | 26.3 (20.5) [20.5 to 32.7]
  Redness: Moderate | 20.0 (15.0) [15.0 to 25.8] | 23.7 (18.3) [18.3 to 29.8] | 11.1 (7.2) [7.2 to 16.0]
  Redness: Severe | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.7]
  Swelling: Mild | 48.9 (42.2) [42.2 to 55.6] | 42.9 (36.3) [36.3 to 49.6] | 17.5 (12.7) [12.7 to 23.2]
  Swelling: Moderate | 19.6 (14.6) [14.6 to 25.3] | 23.2 (17.9) [17.9 to 29.3] | 11.1 (7.2) [7.2 to 16.0]
  Swelling: Severe | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.7]
  Pain at the injection site: Mild | 15.6 (11.1) [11.1 to 21.0] | 13.4 (9.2) [9.2 to 18.6] | 12.4 (8.4) [8.4 to 17.6]
  Pain at the injection site: Moderate | 1.8 (0.5) [0.5 to 4.5] | 2.7 (1.0) [1.0 to 5.7] | 3.2 (1.3) [1.3 to 6.5]
  Pain at the injection site: Severe | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.6] | 0.5 (0.0) [0.0 to 2.5]

2. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 2
Description: Local reactions included pain at injection site, redness and swelling were measured and recorded in measuring device (caliper) units. 1 measuring device unit =0.5 cm. Pain at injection site was graded as mild: hurts if gently touched; moderate: hurts if gently touched with crying; severe: limited limb movement. Redness and swelling were graded as mild: >0 to 2.0 cm; moderate >2.0 to 7.0 cm; and severe: >7.0 cm.
Time Frame: Within 7 Days after Dose 2
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after Dose 2. Here, "Number of Participants Analyzed" = number of participants with any e-diary data reported after Dose 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 223 | 222 | 215
Percentage of participants
  Redness: Mild | 52.9 (46.1) [46.1 to 59.6] | 53.2 (46.4) [46.4 to 59.9] | 24.7 (19.0) [19.0 to 31.0]
  Redness: Moderate | 23.3 (17.9) [17.9 to 29.4] | 31.1 (25.1) [25.1 to 37.6] | 7.0 (4.0) [4.0 to 11.2]
  Redness: Severe | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.7]
  Swelling: Mild | 46.2 (39.5) [39.5 to 53.0] | 46.8 (40.1) [40.1 to 53.6] | 18.1 (13.2) [13.2 to 24.0]
  Swelling: Moderate | 22.4 (17.1) [17.1 to 28.5] | 26.6 (20.9) [20.9 to 32.9] | 7.9 (4.7) [4.7 to 12.4]
  Swelling: Severe | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.7]
  Pain at the injection site: Mild | 13.0 (8.9) [8.9 to 18.1] | 16.7 (12.0) [12.0 to 22.2] | 9.3 (5.8) [5.8 to 14.0]
  Pain at the injection site: Moderate | 3.6 (1.6) [1.6 to 6.9] | 0.5 (0.0) [0.0 to 2.5] | 2.3 (0.8) [0.8 to 5.3]
  Pain at the injection site: Severe | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.7]

3. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 3
Description: as for outcome 2
Time Frame: Within 7 Days after Dose 3
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after Dose 3. Here, "Overall Number of Participants Analyzed" = number of participants with any e-diary data reported after Dose 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 222 | 221 | 215
Percentage of participants
  Redness: Mild | 45.0 [38.4 to 51.8] | 51.1 [44.3 to 57.9] | 23.3 [17.8 to 29.5]
  Redness: Moderate | 33.8 [27.6 to 40.4] | 34.8 [28.6 to 41.5] | 8.4 [5.0 to 12.9]
  Redness: Severe | 0 [0.0 to 1.6] | 0 [0.0 to 1.7] | 0 [0.0 to 1.7]
  Swelling: Mild | 38.7 [32.3 to 45.5] | 39.8 [33.3 to 46.6] | 17.7 [12.8 to 23.4]
  Swelling: Moderate | 30.2 [24.2 to 36.7] | 35.3 [29.0 to 42.0] | 9.8 [6.1 to 14.5]
  Swelling: Severe | 0 [0.0 to 1.6] | 0 [0.0 to 1.7] | 0 [0.0 to 1.7]
  Pain at the injection site: Mild | 10.8 [7.1 to 15.7] | 14.5 [10.1 to 19.8] | 8.8 [5.4 to 13.5]
  Pain at the injection site: Moderate | 3.6 [1.6 to 7.0] | 1.4 [0.3 to 3.9] | 0.9 [0.1 to 3.3]
  Pain at the injection site: Severe | 0 [0.0 to 1.6] | 0 [0.0 to 1.7] | 0.5 [0.0 to 2.6]

4. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 4
Description: as for outcome 2
Time Frame: Within 7 Days after Dose 4
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after Dose 4. Here, "Number of Participants Analyzed" = number of participants with any e-diary data reported after Dose 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 218 | 220 | 212
Percentage of participants
  Redness: Mild | 37.2 [30.7 to 43.9] | 36.4 [30.0 to 43.1] | 20.8 [15.5 to 26.8]
  Redness: Moderate | 49.1 [42.3 to 55.9] | 49.1 [42.3 to 55.9] | 11.8 [7.8 to 16.9]
  Redness: Severe | 0.5 [0.0 to 2.5] | 0.5 [0.0 to 2.5] | 0 [0.0 to 1.7]
  Swelling: Mild | 37.6 [31.2 to 44.4] | 35.9 [29.6 to 42.6] | 13.2 [9.0 to 18.5]
  Swelling: Moderate | 42.2 [35.6 to 49.1] | 41.8 [35.2 to 48.6] | 10.8 [7.0 to 15.8]
  Swelling: Severe | 0.5 [0.0 to 2.5] | 0 [0.0 to 1.7] | 0 [0.0 to 1.7]
  Pain at the injection site: Mild | 19.7 [14.7 to 25.6] | 19.1 [14.1 to 24.9] | 10.4 [6.6 to 15.3]
  Pain at the injection site: Moderate | 1.4 [0.3 to 4.0] | 3.2 [1.3 to 6.4] | 3.3 [1.3 to 6.7]
  Pain at the injection site: Severe | 0 [0.0 to 1.7] | 0 [0.0 to 1.7] | 0 [0.0 to 1.7]

5. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 1
Description: Systemic events included fever, decreased appetite, drowsiness and irritability. Fever was defined as an axillary temperature greater than or equal to (>=) 37.5 degree Celsius (C), and categorized as >=37.5 to 38.4 degree C, greater than (>)38.4 to 38.9 degree C,>38.9 to 40.0 degree C and >40.0 degree C; decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed); drowsiness was graded as mild (increased or prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity); Irritability: graded as mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted).
Time Frame: Within 7 Days After Dose 1
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up Dose 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 225 | 224 | 217
Percentage of participants
  Fever: >=37.5 degree C | 9.8 (6.2) [6.2 to 14.4] | 12.9 (8.8) [8.8 to 18.1] | 9.7 (6.1) [6.1 to 14.4]
  Fever: >=37.5°C to 38.4 degree C | 9.3 (5.9) [5.9 to 13.9] | 12.5 (8.5) [8.5 to 17.6] | 9.7 (6.1) [6.1 to 14.4]
  Fever: >38.4°C to 38.9 degree C | 0.4 (0.0) [0.0 to 2.5] | 0.4 (0.0) [0.0 to 2.5] | 0 (0.0) [0.0 to 1.7]
  Fever: >38.9 to 40.0 degree C | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.7]
  Fever: >40.0 degree C | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.7]
  Decreased appetite: Mild | 3.6 (1.5) [1.5 to 6.9] | 7.1 (4.1) [4.1 to 11.3] | 3.2 (1.3) [1.3 to 6.5]
  Decreased appetite: Moderate | 1.8 (0.5) [0.5 to 4.5] | 3.1 (1.3) [1.3 to 6.3] | 3.2 (1.3) [1.3 to 6.5]
  Decreased appetite: Severe | 0 (0.0) [0.0 to 1.6] | 0.4 (0.0) [0.0 to 2.5] | 0 (0.0) [0.0 to 1.7]
  Drowsiness: Mild | 40.4 (34.0) [34.0 to 47.2] | 42.0 (35.4) [35.4 to 48.7] | 42.9 (36.2) [36.2 to 49.7]
  Drowsiness: Moderate | 0.9 (0.1) [0.1 to 3.2] | 2.2 (0.7) [0.7 to 5.1] | 4.1 (1.9) [1.9 to 7.7]
  Drowsiness: Severe | 0 (0.0) [0.0 to 1.6] | 0.4 (0.0) [0.0 to 2.5] | 0 (0.0) [0.0 to 1.7]
  Irritability: Mild | 13.8 (9.6) [9.6 to 19.0] | 11.2 (7.4) [7.4 to 16.0] | 12.9 (8.7) [8.7 to 18.1]
  Irritability: Moderate | 12.0 (8.1) [8.1 to 17.0] | 13.4 (9.2) [9.2 to 18.6] | 11.5 (7.6) [7.6 to 16.5]
  Irritability: Severe | 1.3 (0.3) [0.3 to 3.8] | 1.8 (0.5) [0.5 to 4.5] | 0.5 (0.0) [0.0 to 2.5]

6. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 2
Description: Systemic events included fever, decreased appetite, drowsiness and irritability. Fever was defined as an axillary temperature >=37.5 degree C and categorized as >=37.5 to 38.4 degree C,>38.4 to 38.9 degree C,>38.9 to 40.0 degree C and >40.0 degree C; decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed); drowsiness was graded as mild (increased or prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity); Irritability: graded as mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted).
Time Frame: Within 7 Days After Dose 2
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after Dose 2. Here, "Overall Number of Participants Analyzed" = number of participants with any e-diary data reported after Dose 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 223 | 222 | 215
Percentage of participants
  Fever: >=37.5 degree C | 20.2 (15.1) [15.1 to 26.1] | 21.2 (16.0) [16.0 to 27.1] | 18.1 (13.2) [13.2 to 24.0]
  Fever: >=37.5 to 38.4 degree C | 15.2 (10.8) [10.8 to 20.6] | 17.6 (12.8) [12.8 to 23.2] | 14.9 (10.4) [10.4 to 20.4]
  Fever: >38.4 to 38.9 degree C | 3.1 (1.3) [1.3 to 6.4] | 2.3 (0.7) [0.7 to 5.2] | 1.9 (0.5) [0.5 to 4.7]
  Fever: >38.9 to 40.0 degree C | 1.8 (0.5) [0.5 to 4.5] | 1.4 (0.3) [0.3 to 3.9] | 1.4 (0.3) [0.3 to 4.0]
  Fever: >40.0 degree C | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.7]
  Decreased appetite: Mild | 4.5 (2.2) [2.2 to 8.1] | 6.8 (3.8) [3.8 to 10.9] | 5.1 (2.6) [2.6 to 9.0]
  Decreased appetite: Moderate | 5.8 (3.1) [3.1 to 9.8] | 5.0 (2.5) [2.5 to 8.7] | 4.7 (2.3) [2.3 to 8.4]
  Decreased appetite: Severe | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.7]
  Drowsiness: Mild | 39.9 (33.4) [33.4 to 46.7] | 48.6 (41.9) [41.9 to 55.4] | 39.5 (33.0) [33.0 to 46.4]
  Drowsiness: Moderate | 3.1 (1.3) [1.3 to 6.4] | 4.1 (1.9) [1.9 to 7.6] | 2.3 (0.8) [0.8 to 5.3]
  Drowsiness: Severe | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.7]
  Irritability: Mild | 12.6 (8.5) [8.5 to 17.6] | 16.7 (12.0) [12.0 to 22.2] | 10.2 (6.5) [6.5 to 15.1]
  Irritability: Moderate | 12.1 (8.1) [8.1 to 17.1] | 14.9 (10.5) [10.5 to 20.2] | 15.3 (10.8) [10.8 to 20.9]
  Irritability: Severe | 1.3 (0.3) [0.3 to 3.9] | 0.5 (0.0) [0.0 to 2.5] | 1.4 (0.3) [0.3 to 4.0]

7. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 3
Description: as for outcome 6
Time Frame: Within 7 Days After Dose 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 222 | 221 | 215
Percentage of participants
  Fever: >=37.5 degree C | 15.3 (10.8) [10.8 to 20.7] | 19.9 (14.9) [14.9 to 25.8] | 15.3 (10.8) [10.8 to 20.9]
  Fever: >=37.5 to 38.4 degree C | 13.5 (9.3) [9.3 to 18.7] | 16.3 (11.7) [11.7 to 21.8] | 12.6 (8.4) [8.4 to 17.7]
  Fever: >38.4 to 38.9 degree C | 1.4 (0.3) [0.3 to 3.9] | 2.7 (1.0) [1.0 to 5.8] | 1.9 (0.5) [0.5 to 4.7]
  Fever: >38.9 to 40.0 degree C | 0.5 (0.0) [0.0 to 2.5] | 0.9 (0.1) [0.1 to 3.2] | 0.9 (0.1) [0.1 to 3.3]
  Fever: >40.0 degree C | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.7] | 0 (0.0) [0.0 to 1.7]
  Decreased appetite: Mild | 5.0 (2.5) [2.5 to 8.7] | 7.2 (4.2) [4.2 to 11.5] | 4.2 (1.9) [1.9 to 7.8]
  Decreased appetite: Moderate | 2.7 (1.0) [1.0 to 5.8] | 3.6 (1.6) [1.6 to 7.0] | 3.7 (1.6) [1.6 to 7.2]
  Decreased appetite: Severe | 0.5 (0.0) [0.0 to 2.5] | 0 (0.0) [0.0 to 1.7] | 0 (0.0) [0.0 to 1.7]
  Drowsiness: Mild | 24.8 (19.2) [19.2 to 31.0] | 32.6 (26.4) [26.4 to 39.2] | 32.6 (26.3) [26.3 to 39.3]
  Drowsiness: Moderate | 1.4 (0.3) [0.3 to 3.9] | 1.8 (0.5) [0.5 to 4.6] | 1.4 (0.3) [0.3 to 4.0]
  Drowsiness: Severe | 0 (0.0) [0.0 to 1.6] | 0 (0.0) [0.0 to 1.7] | 0 (0.0) [0.0 to 1.7]
  Irritability: Mild | 16.7 (12.0) [12.0 to 22.2] | 10.9 (7.1) [7.1 to 15.7] | 14.0 (9.6) [9.6 to 19.3]
  Irritability: Moderate | 8.6 (5.2) [5.2 to 13.0] | 9.0 (5.6) [5.6 to 13.6] | 13.0 (8.8) [8.8 to 18.3]
  Irritability: Severe | 0.5 (0.0) [0.0 to 2.5] | 0 (0.0) [0.0 to 1.7] | 0.9 (0.1) [0.1 to 3.3]

8. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 4
Description: as for outcome 6
Time Frame: Within 7 Days After Dose 4
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after Dose 4. Here, "Overall Number of Participants Analyzed" = number of participants with any e-diary data reported after Dose 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 218 | 220 | 212
Percentage of participants
  Fever: >=37.5 degree C | 42.7 (36.0) [36.0 to 49.5] | 39.5 (33.0) [33.0 to 46.3] | 38.2 (31.6) [31.6 to 45.1]
  Fever: >=37.5 to 38.4 degree C | 25.7 (20.0) [20.0 to 32.0] | 29.1 (23.2) [23.2 to 35.6] | 24.1 (18.5) [18.5 to 30.4]
  Fever: >38.4 to 38.9 degree C | 10.1 (6.4) [6.4 to 14.9] | 5.9 (3.2) [3.2 to 9.9] | 6.1 (3.3) [3.3 to 10.3]
  Fever: >38.9 to 40.0 degree C | 6.4 (3.6) [3.6 to 10.5] | 4.5 (2.2) [2.2 to 8.2] | 8.0 (4.7) [4.7 to 12.5]
  Fever: >40.0 degree C | 0.5 (0.0) [0.0 to 2.5] | 0 (0.0) [0.0 to 1.7] | 0 (0.0) [0.0 to 1.7]
  Decreased appetite: Mild | 6.4 (3.6) [3.6 to 10.5] | 6.8 (3.9) [3.9 to 11.0] | 6.1 (3.3) [3.3 to 10.3]
  Decreased appetite: Moderate | 7.3 (4.3) [4.3 to 11.6] | 7.7 (4.6) [4.6 to 12.1] | 5.7 (3.0) [3.0 to 9.7]
  Decreased appetite: Severe | 0 (0.0) [0.0 to 1.7] | 0 (0.0) [0.0 to 1.7] | 0.9 (0.1) [0.1 to 3.4]
  Drowsiness: Mild | 24.3 (18.8) [18.8 to 30.6] | 23.6 (18.2) [18.2 to 29.8] | 29.7 (23.7) [23.7 to 36.4]
  Drowsiness: Moderate | 1.4 (0.3) [0.3 to 4.0] | 2.3 (0.7) [0.7 to 5.2] | 1.9 (0.5) [0.5 to 4.8]
  Drowsiness: Severe | 0 (0.0) [0.0 to 1.7] | 0 (0.0) [0.0 to 1.7] | 0 (0.0) [0.0 to 1.7]
  Irritability: Mild | 14.2 (9.9) [9.9 to 19.6] | 15.5 (10.9) [10.9 to 20.9] | 15.1 (10.6) [10.6 to 20.6]
  Irritability: Moderate | 7.3 (4.3) [4.3 to 11.6] | 11.4 (7.5) [7.5 to 16.3] | 9.4 (5.9) [5.9 to 14.2]
  Irritability: Severe | 0.9 (0.1) [0.1 to 3.3] | 0.9 (0.1) [0.1 to 3.2] | 0.5 (0.0) [0.0 to 2.6]

9. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Dose 1 to 1 Month After Dose 3
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Day 1 of Dose 1 to 1 Month after Dose 3
Population: Safety population included all the participants who received at least 1 dose of the IP and had safety data after any dose.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 225 | 224 | 217
Percentage of participants | 47.6 (40.9) [40.9 to 54.3] | 55.4 (48.6) [48.6 to 62.0] | 58.5 (51.7) [51.7 to 65.2]

10. Primary Outcome: Percentage of Participants With AEs From Dose 4 to 1 Month After Dose 4
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: From Dose 4 to 1 Month after Dose 4
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after any dose. Here, "Number of Participants Analyzed" = number of participants who received Dose 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 218 | 220 | 212
Percentage of participants | 40.4 (33.8) [33.8 to 47.2] | 43.2 (36.5) [36.5 to 50.0] | 43.9 (37.1) [37.1 to 50.8]

11. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) From Dose 1 to 1 Month After Dose 4
Description: A serious AE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect and other important medical events.
Time Frame: From Dose 1 to 1 Month after Dose 4
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after any dose.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 225 | 224 | 217
Percentage of participants | 6.2 (3.4) [3.4 to 10.2] | 4.0 (1.9) [1.9 to 7.5] | 7.4 (4.3) [4.3 to 11.7]

12. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) From Dose 1 to 1 Month After Dose 4
Description: An NDCMC was defined as a significant disease or medical condition, not previously identified, that is expected to be persistent or was otherwise long-lasting in its effects.
Time Frame: From Dose 1 to 1 Month after Dose 4
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after any dose. Here, "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 225 | 224 | 217
Percentage of participants | 10.7 (7.0) [7.0 to 15.5] | 8.9 (5.5) [5.5 to 13.5] | 8.3 (5.0) [5.0 to 12.8]

13. Primary Outcome: Percentage of Participants With Predefined Pneumococcal Serotype-specific Immunoglobulin G (IgG) Concentrations 1 Month After Dose 3
Description: Pneumococcal serotype-specific IgG Concentrations were measured for 20vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F. Assay results below the lower limit of quantitation (LLOQ) were set to 0.5*LLOQ. The predefined levels, >=0.35 micrograms/mL for all serotypes except for serotypes 5 (>=0.23 micrograms/mL), 6B (>=0.10 micrograms/mL) and 19A (>=0.12 micrograms/mL).
Time Frame: 1 Month after Dose 3
Population: Dose 3 evaluable immunogenicity population included eligible participants who were 2 to 6 months of age at first vaccination, received first 3 doses as randomized, had at least 1 valid immunogenicity results from blood collection within 27 to 56 days after Dose 3, had no other major protocol deviations per clinician.Here, "N" = participants with an IgG concentration greater than or equal to(>=)predefined level for given serotype,"n" =participants with valid assay results for specified serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 221 | 220 | 213
Percentage of participants
  Serotype: 1 | 97.7 [94.8 to 99.3] | 99.1 [96.8 to 99.9] | 92.0 [87.5 to 95.3]
  Serotype: 3 | 96.4 [93.0 to 98.4] | 99.1 [96.8 to 99.9] | 95.3 [91.5 to 97.7]
  Serotype: 4 | 96.8 [93.6 to 98.7] | 99.1 [96.8 to 99.9] | 94.8 [90.9 to 97.4]
  Serotype: 5 | 92.3 [88.0 to 95.5] | 97.3 [94.2 to 99.0] | 93.0 [88.7 to 96.0]
  Serotype: 6A | 90.0 [85.3 to 93.7] | 98.2 [95.4 to 99.5] | 94.8 [90.9 to 97.4]
  Serotype: 6B | 87.8 [82.7 to 91.8] | 96.4 [93.0 to 98.4] | 82.2 [76.3 to 87.1]
  Serotype: 7F | 95.9 [92.4 to 98.1] | 99.1 [96.8 to 99.9] | 94.8 [90.9 to 97.4]
  Serotype: 9V | 95.9 [92.4 to 98.1] | 98.6 [96.1 to 99.7] | 93.0 [88.7 to 96.0]
  Serotype: 14: number analyzed (Participants) | 220 | 220 | 213
  Serotype: 14 | 96.8 [93.6 to 98.7] | 97.7 [94.8 to 99.3] | 96.2 [92.7 to 98.4]
  Serotype: 18C | 96.8 [93.6 to 98.7] | 99.1 [96.8 to 99.9] | 94.8 [90.9 to 97.4]
  Serotype: 19A | 99.5 [97.5 to 100.0] | 99.5 [97.5 to 100.0] | 99.1 [96.6 to 99.9]
  Serotype: 19F | 100.0 [98.3 to 100.0] | 100.0 [98.3 to 100.0] | 100.0 [98.3 to 100.0]
  Serotype: 23F | 89.6 [84.8 to 93.3] | 93.6 [89.6 to 96.5] | 88.7 [83.7 to 92.6]
  Serotype: 8: number analyzed (Participants) | 221 | 219 | 213
  Serotype: 8 | 99.5 [97.5 to 100.0] | 0.9 [0.1 to 3.3] | 99.5 [97.4 to 100.0]
  Serotype: 10A | 60.2 [53.4 to 66.7] | 1.8 [0.5 to 4.6] | 59.6 [52.7 to 66.3]
  Serotype: 11A | 100.0 [98.3 to 100.0] | 2.7 [1.0 to 5.8] | 100.0 [98.3 to 100.0]
  Serotype: 12F | 74.7 [68.4 to 80.3] | 0.9 [0.1 to 3.2] | 74.6 [68.3 to 80.3]
  Serotype: 15B | 99.1 [96.8 to 99.9] | 8.2 [4.9 to 12.6] | 98.6 [95.9 to 99.7]
  Serotype: 22F | 100.0 [98.3 to 100.0] | 0.9 [0.1 to 3.2] | 100.0 [98.3 to 100.0]
  Serotype: 33F: number analyzed (Participants) | 219 | 220 | 212
  Serotype: 33F | 95.0 [91.2 to 97.5] | 3.2 [1.3 to 6.4] | 92.5 [88.0 to 95.6]
Statistical Analysis 1: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 1: 2-Sided 95% CIs are calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC (SC) is to the corresponding serotype in 13vPnC (SC) group. Noninferiority was declared if the lower bound of the 2-sided 95% CIs for the percentage differences (20vPnC SC - 13vPnC SC) was greater than -10%; Percentage Difference = -1.4, 95% CI 2-sided [-4.4 to 1.3]
Statistical Analysis 2: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 3: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Percentage Difference = -2.7, 95% CI 2-sided [-6.2 to 0.1]
Statistical Analysis 3: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 4: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Percentage Difference = -2.3, 95% CI 2-sided [-5.6 to 0.5]
Statistical Analysis 4: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 5: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Percentage Difference = -5.0, 95% CI 2-sided [-9.6 to -0.9]
Statistical Analysis 5: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 6A: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Percentage Difference = -8.1, 95% CI 2-sided [-13.0 to -4.0]
Statistical Analysis 6: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 6B: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Percentage Difference = -8.6, 95% CI 2-sided [-14.0 to -3.7]
Statistical Analysis 7: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 7F: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Percentage Difference = -3.2, 95% CI 2-sided [-6.8 to -0.3]
Statistical Analysis 8: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 9V: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Percentage Difference = -2.7, 95% CI 2-sided [-6.4 to 0.4]
Statistical Analysis 9: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 14: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Percentage Difference = -0.9, 95% CI 2-sided [-4.4 to 2.4]
Statistical Analysis 10: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 18C: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Percentage Difference = -2.3, 95% CI 2-sided [-5.6 to 0.5]
Statistical Analysis 11: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 19A: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Percentage Difference = 0.0, 95% CI 2-sided [-2.1 to 2.1]
Statistical Analysis 12: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 19F: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Percentage Difference = 0.0, 95% CI 2-sided [-1.7 to 1.7]
Statistical Analysis 13: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 23F: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Percentage Difference = -4.0, 95% CI 2-sided [-9.5 to 1.2]
Statistical Analysis 14: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 8: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — For the additional 7 serotypes, the compared results are from serotype 23F (13vPnC [SC] serotype with the lowest percentage, not including serotype 3) in the 13vPnC (SC) group. Noninferiority was declared if the lower bound of the 2-sided 95% CIs for the percentage differences (20vPnC SC - lowest 13vPnC SC) was greater than -10%; Percentage Difference = 5.9, 95% CI 2-sided [3.0 to 10.0]
Statistical Analysis 15: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 10A: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; Percentage Difference = -33.5, 95% CI 2-sided [-40.7 to -26.2]
Statistical Analysis 16: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 11A: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; Percentage Difference = 6.4, 95% CI 2-sided [3.8 to 10.4]
Statistical Analysis 17: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 12F: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; Percentage Difference = -19.0, 95% CI 2-sided [-25.7 to -12.5]
Statistical Analysis 18: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 15B: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; Percentage Difference = 5.5, 95% CI 2-sided [2.2 to 9.6]
Statistical Analysis 19: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 22F: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; Percentage Difference = 6.4, 95% CI 2-sided [3.8 to 10.4]
Statistical Analysis 20: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 33F: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; Percentage Difference = 1.3, 95% CI 2-sided [-3.2 to 6.0]
Statistical Analysis 21: Comparison: 20vPnC (SC) vs 20vPnC (IM); Serotype 1: 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage; Test type: Other; Percentage Difference = -5.7, 95% CI 2-sided [-10.4 to -1.7]
Statistical Analysis 22: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 2]; Test type: Other; Percentage Difference = -1.1, 95% CI 2-sided [-5.2 to 2.9]
Statistical Analysis 23: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 3]; Test type: Other; Percentage Difference = -2.0, 95% CI 2-sided [-6.2 to 1.9]
Statistical Analysis 24: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 4]; Test type: Other; Percentage Difference = 0.7, 95% CI 2-sided [-4.5 to 5.8]
Statistical Analysis 25: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 5]; Test type: Other; Percentage Difference = 4.8, 95% CI 2-sided [-0.2 to 10.0]
Statistical Analysis 26: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 6]; Test type: Other; Percentage Difference = -5.6, 95% CI 2-sided [-12.5 to 1.1]
Statistical Analysis 27: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 7]; Test type: Other; Percentage Difference = -1.1, 95% CI 2-sided [-5.4 to 3.1]
Statistical Analysis 28: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 8]; Test type: Other; Percentage Difference = -3.0, 95% CI 2-sided [-7.7 to 1.4]
Statistical Analysis 29: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 9]; Test type: Other; Percentage Difference = -0.6, 95% CI 2-sided [-4.4 to 3.2]
Statistical Analysis 30: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 10]; Test type: Other; Percentage Difference = -2.0, 95% CI 2-sided [-6.2 to 1.9]
Statistical Analysis 31: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 11]; Test type: Other; Percentage Difference = -0.5, 95% CI 2-sided [-3.0 to 1.7]
Statistical Analysis 32: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 12]; Test type: Other; Percentage Difference = 0.0, 95% CI 2-sided [-1.8 to 1.7]
Statistical Analysis 33: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 13]; Test type: Other; Percentage Difference = -0.9, 95% CI 2-sided [-6.9 to 5.1]
Statistical Analysis 34: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 14]; Test type: Other; Percentage Difference = 0.0, 95% CI 2-sided [-2.2 to 2.1]
Statistical Analysis 35: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 15]; Test type: Other; Percentage Difference = -0.6, 95% CI 2-sided [-9.8 to 8.6]
Statistical Analysis 36: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 16]; Test type: Other; Percentage Difference = 0.0, 95% CI 2-sided [-1.8 to 1.7]
Statistical Analysis 37: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 17]; Test type: Other; Percentage Difference = 0.0, 95% CI 2-sided [-8.2 to 8.2]
Statistical Analysis 38: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 18]; Test type: Other; Percentage Difference = -0.5, 95% CI 2-sided [-3.3 to 2.0]
Statistical Analysis 39: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 19]; Test type: Other; Percentage Difference = 0.0, 95% CI 2-sided [-1.8 to 1.7]
Statistical Analysis 40: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 13, analysis 20]; Test type: Other; Percentage Difference = -2.5, 95% CI 2-sided [-7.5 to 2.2]

14. Secondary Outcome: Geometric Mean Concentration of Pneumococcal Serotype-Specific IgG Concentrations 1 Month After Dose 3
Description: Pneumococcal serotype-specific IgG concentrations were measured for 20vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F. Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: 1 Month after Dose 3
Population: Dose 3 evaluable immunogenicity population included eligible participants who were 2 to 6 months of age at first vaccination, received first 3 doses as randomized, had at least 1 valid immunogenicity results from blood collection within 27 to 56 days after Dose 3, and had no other major protocol deviations per clinician. Here, "N" = participants with an IgG concentration >= predefined level for given serotype and "n" =participants with valid assay results for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 221 | 220 | 213
Micrograms per milliliter
  Serotype 1 | 1.37 [1.25 to 1.51] | 2.21 [1.98 to 2.47] | 1.17 [1.04 to 1.31]
  Serotype 3 | 1.29 [1.18 to 1.41] | 1.81 [1.66 to 1.98] | 1.10 [0.99 to 1.22]
  Serotype 4 | 1.76 [1.57 to 1.97] | 2.96 [2.64 to 3.32] | 1.73 [1.52 to 1.97]
  Serotype 5 | 1.01 [0.89 to 1.16] | 1.72 [1.51 to 1.96] | 1.00 [0.87 to 1.14]
  Serotype 6A | 1.38 [1.21 to 1.57] | 2.34 [2.09 to 2.62] | 1.64 [1.42 to 1.88]
  Serotype 6B | 0.42 [0.35 to 0.50] | 0.83 [0.71 to 0.97] | 0.39 [0.32 to 0.48]
  Serotype 7F | 1.58 [1.43 to 1.75] | 2.19 [1.95 to 2.46] | 1.52 [1.35 to 1.71]
  Serotype 9V | 1.46 [1.32 to 1.61] | 2.11 [1.88 to 2.36] | 1.45 [1.29 to 1.64]
  Serotype 14: number analyzed (Participants) | 220 | 220 | 213
  Serotype 14 | 2.79 [2.45 to 3.18] | 3.31 [2.90 to 3.78] | 2.43 [2.13 to 2.76]
  Serotype 18C | 1.67 [1.51 to 1.86] | 2.52 [2.26 to 2.82] | 1.54 [1.38 to 1.72]
  Serotype 19A | 2.41 [2.19 to 2.65] | 3.19 [2.86 to 3.56] | 2.36 [2.11 to 2.64]
  Serotype 19F | 2.81 [2.60 to 3.04] | 3.73 [3.41 to 4.08] | 2.76 [2.53 to 3.02]
  Serotype 23F | 1.32 [1.15 to 1.51] | 2.05 [1.79 to 2.34] | 1.29 [1.13 to 1.48]
  Serotype 8: number analyzed (Participants) | 221 | 219 | 213
  Serotype 8 | 3.32 [3.05 to 3.61] | 0.01 [0.01 to 0.01] | 3.29 [2.97 to 3.64]
  Serotype 10A | 0.50 [0.42 to 0.60] | 0.01 [0.01 to 0.02] | 0.47 [0.39 to 0.56]
  Serotype 11A | 5.63 [5.17 to 6.14] | 0.02 [0.02 to 0.02] | 5.22 [4.73 to 5.77]
  Serotype 12F | 0.79 [0.67 to 0.93] | 0.01 [0.01 to 0.01] | 0.72 [0.60 to 0.85]
  Serotype 15B | 6.77 [6.04 to 7.60] | 0.04 [0.03 to 0.05] | 6.80 [6.03 to 7.67]
  Serotype 22F | 4.94 [4.54 to 5.38] | 0.01 [0.00 to 0.01] | 4.41 [3.99 to 4.88]
  Serotype 33F: number analyzed (Participants) | 219 | 220 | 212
  Serotype 33F | 1.70 [1.51 to 1.92] | 0.02 [0.02 to 0.03] | 1.62 [1.40 to 1.87]
Statistical Analysis 1: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 1: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC (SC) is to the corresponding serotype in 13vPnC (SC) group. Noninferiority was declared if the lower bound of the 2-sided 95% CI for the GMR (20vPnC [SC]/13vPnC [SC]) was greater than 0.5 (2-fold criterion); GMR = 0.62, 95% CI 2-sided [0.54 to 0.72]
Statistical Analysis 2: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 3: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; GMR = 0.71, 95% CI 2-sided [0.63 to 0.81]
Statistical Analysis 3: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 4: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; GMR = 0.60, 95% CI 2-sided [0.51 to 0.70]
Statistical Analysis 4: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 5: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; GMR = 0.59, 95% CI 2-sided [0.49 to 0.71]
Statistical Analysis 5: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 6A: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; GMR = 0.59, 95% CI 2-sided [0.50 to 0.70]
Statistical Analysis 6: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 6B: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; GMR = 0.51, 95% CI 2-sided [0.40 to 0.64]
Statistical Analysis 7: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 7F: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; GMR = 0.72, 95% CI 2-sided [0.62 to 0.84]
Statistical Analysis 8: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 9V: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; GMR = 0.69, 95% CI 2-sided [0.60 to 0.80]
Statistical Analysis 9: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 14: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; GMR = 0.84, 95% CI 2-sided [0.70 to 1.01]
Statistical Analysis 10: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 18C: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; GMR = 0.66, 95% CI 2-sided [0.57 to 0.77]
Statistical Analysis 11: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 19A: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; GMR = 0.76, 95% CI 2-sided [0.65 to 0.87]
Statistical Analysis 12: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 19F: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; GMR = 0.75, 95% CI 2-sided [0.67 to 0.85]
Statistical Analysis 13: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 23F: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; GMR = 0.64, 95% CI 2-sided [0.53 to 0.78]
Statistical Analysis 14: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 8: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — For the additional 7 serotypes, the compared results are from serotype 6B (13vPnC [SC] serotype with the lowest GMC, not including serotype 3) in the 13vPnC (SC) group. Noninferiority was declared if the lower bound of the 2-sided 95% CI for the GMR (20vPnC [SC]/lowest 13vPnC [SC]) was greater than 0.5 (2-fold criterion); GMR = 4.01, 95% CI 2-sided [3.36 to 4.79]
Statistical Analysis 15: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 10A: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 14]; GMR = 0.60, 95% CI 2-sided [0.48 to 0.76]
Statistical Analysis 16: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 11A: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 14]; GMR = 6.80, 95% CI 2-sided [5.69 to 8.13]
Statistical Analysis 17: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 12F: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 14]; GMR = 0.95, 95% CI 2-sided [0.76 to 1.20]
Statistical Analysis 18: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 15B: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 14]; GMR = 8.18, 95% CI 2-sided [6.75 to 9.92]
Statistical Analysis 19: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 22F: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 14]; GMR = 5.97, 95% CI 2-sided [5.00 to 7.12]
Statistical Analysis 20: Comparison: 20vPnC (SC) vs 13vPnC (SC); Serotype 33F: 2-Sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the IgG concentrations and the corresponding CIs based on the geometric mean ratio; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 14]; GMR = 2.06, 95% CI 2-sided [1.69 to 2.51]
Statistical Analysis 21: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 1]; Test type: Other; GMR = 0.85, 95% CI 2-sided [0.73 to 0.99]
Statistical Analysis 22: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 2]; Test type: Other; GMR = 0.85, 95% CI 2-sided [0.74 to 0.98]
Statistical Analysis 23: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 3]; Test type: Other; GMR = 0.98, 95% CI 2-sided [0.83 to 1.16]
Statistical Analysis 24: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 4]; Test type: Other; GMR = 0.98, 95% CI 2-sided [0.81 to 1.19]
Statistical Analysis 25: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 5]; Test type: Other; GMR = 1.19, 95% CI 2-sided [0.98 to 1.44]
Statistical Analysis 26: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 6]; Test type: Other; GMR = 0.93, 95% CI 2-sided [0.72 to 1.21]
Statistical Analysis 27: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 7]; Test type: Other; GMR = 0.96, 95% CI 2-sided [0.82 to 1.12]
Statistical Analysis 28: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 8]; Test type: Other; GMR = 0.99, 95% CI 2-sided [0.85 to 1.16]
Statistical Analysis 29: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 9]; Test type: Other; GMR = 0.87, 95% CI 2-sided [0.72 to 1.04]
Statistical Analysis 30: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 10]; Test type: Other; GMR = 0.92, 95% CI 2-sided [0.79 to 1.07]
Statistical Analysis 31: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 11]; Test type: Other; GMR = 0.98, 95% CI 2-sided [0.84 to 1.13]
Statistical Analysis 32: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 12]; Test type: Other; GMR = 0.98, 95% CI 2-sided [0.87 to 1.10]
Statistical Analysis 33: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 13]; Test type: Other; GMR = 0.98, 95% CI 2-sided [0.81 to 1.19]
Statistical Analysis 34: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 14]; Test type: Other; GMR = 0.99, 95% CI 2-sided [0.87 to 1.13]
Statistical Analysis 35: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 15]; Test type: Other; GMR = 0.94, 95% CI 2-sided [0.73 to 1.20]
Statistical Analysis 36: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 16]; Test type: Other; GMR = 0.93, 95% CI 2-sided [0.81 to 1.06]
Statistical Analysis 37: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 17]; Test type: Other; GMR = 0.91, 95% CI 2-sided [0.71 to 1.15]
Statistical Analysis 38: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 18]; Test type: Other; GMR = 1.00, 95% CI 2-sided [0.85 to 1.18]
Statistical Analysis 39: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 19]; Test type: Other; GMR = 0.89, 95% CI 2-sided [0.78 to 1.02]
Statistical Analysis 40: Comparison: 20vPnC (SC) vs 20vPnC (IM); [analysis description as in outcome 14, analysis 20]; Test type: Other; GMR = 0.95, 95% CI 2-sided [0.79 to 1.15]

15. Secondary Outcome: Geometric Mean Concentration of Pneumococcal Serotype-Specific IgG Concentrations 1 Month After Dose 4
Description: Pneumococcal serotype-specific IgG concentrations were measured for 20vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F.
Time Frame: 1 Month after Dose 4
Population: Dose 4 evaluable immunogenicity population included eligible participants who were 2 to 6 months of age at Dose 1 and 12 to 15 months of age at Dose 4, received all 4 doses as randomized, had at least 1 valid assay result from the blood collection within 27 to 56 days after Dose 4, and had no other major protocol deviations per clinician. Here,"N" = participants with an IgG concentration >= predefined level for given serotype and "n"=participants with valid assay results for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 217 | 220 | 211
Micrograms per milliliter
  Serotype 1 | 2.79 [2.50 to 3.12] | 4.62 [4.11 to 5.19] | 2.78 [2.47 to 3.12]
  Serotype 3 | 0.97 [0.87 to 1.08] | 1.44 [1.30 to 1.59] | 1.08 [0.96 to 1.21]
  Serotype 4 | 6.93 [6.14 to 7.83] | 10.01 [8.89 to 11.27] | 7.31 [6.51 to 8.20]
  Serotype 5 | 2.96 [2.63 to 3.34] | 4.64 [4.13 to 5.21] | 2.94 [2.59 to 3.33]
  Serotype 6A | 11.90 [10.61 to 13.34] | 17.25 [15.66 to 18.99] | 13.92 [12.43 to 15.59]
  Serotype 6B: number analyzed (Participants) | 216 | 220 | 211
  Serotype 6B | 7.18 [6.30 to 8.18] | 10.48 [9.46 to 11.61] | 7.50 [6.58 to 8.55]
  Serotype 7F | 4.46 [4.04 to 4.92] | 6.62 [5.95 to 7.38] | 4.85 [4.34 to 5.42]
  Serotype 9V | 4.54 [4.04 to 5.09] | 6.62 [5.93 to 7.39] | 5.38 [4.81 to 6.02]
  Serotype 14 | 8.23 [7.27 to 9.31] | 10.30 [9.25 to 11.47] | 9.19 [8.10 to 10.43]
  Serotype 18C | 3.95 [3.50 to 4.45] | 5.97 [5.27 to 6.75] | 3.81 [3.38 to 4.30]
  Serotype 19A: number analyzed (Participants) | 217 | 219 | 211
  Serotype 19A | 7.62 [6.82 to 8.52] | 8.97 [8.08 to 9.95] | 7.92 [7.06 to 8.89]
  Serotype 19F | 8.74 [7.84 to 9.73] | 11.02 [9.96 to 12.20] | 8.56 [7.66 to 9.56]
  Serotype 23F | 7.01 [6.16 to 7.97] | 11.76 [10.42 to 13.28] | 7.39 [6.49 to 8.42]
  Serotype 8: number analyzed (Participants) | 217 | 219 | 211
  Serotype 8 | 5.84 [5.23 to 6.53] | 0.02 [0.02 to 0.03] | 5.88 [5.23 to 6.62]
  Serotype 10A | 6.98 [6.13 to 7.93] | 0.01 [0.01 to 0.01] | 8.02 [7.02 to 9.16]
  Serotype 11A | 5.73 [5.08 to 6.46] | 0.02 [0.01 to 0.02] | 5.78 [5.14 to 6.50]
  Serotype 12F | 2.73 [2.41 to 3.09] | 0.01 [0.01 to 0.01] | 2.69 [2.36 to 3.06]
  Serotype 15B | 18.45 [16.73 to 20.36] | 0.03 [0.03 to 0.04] | 21.83 [19.53 to 24.41]
  Serotype 22F | 14.07 [12.67 to 15.63] | 0.00 [0.00 to 0.01] | 14.21 [12.61 to 16.00]
  Serotype 33F | 10.29 [9.28 to 11.40] | 0.02 [0.01 to 0.02] | 11.13 [9.99 to 12.39]

16. Secondary Outcome: Geometric Mean Titer (GMTs) of Serotype Specific Opsonophagocytic Activity (OPA) at 1 Month After Dose 3, Before Dose 4 and 1 Month After Dose 4
Description: 20vPnC serotypes included: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F. OPA titers were determined in randomly selected subsets of sera from each vaccine group.
Time Frame: 1 Month after Dose 3, before Dose 4 and 1 Month after Dose 4
Population: For 1 month after Dose 3 and before Dose 4: Dose 3 evaluable immunogenicity population set were analyzed and for 1 month after Dose 4: Dose 4 evaluable immunogenicity population for 1 month after Dose 4 OPA GMTs were analyzed. Here, "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure and "Number Analyzed"= participants with valid results for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 73 | 75 | 72
Titers
  Serotype 1:1 Month after Dose 3: number analyzed (Participants) | 71 | 70 | 72
  Serotype 1:1 Month after Dose 3 | 55 [43 to 71] | 126 [104 to 152] | 56 [45 to 70]
  Serotype 1:Before Dose. 4: number analyzed (Participants) | 71 | 71 | 71
  Serotype 1:Before Dose. 4 | 11 [10 to 12] | 13 [11 to 16] | 10 [9 to 11]
  Serotype 1:1 Month after Dose 4: number analyzed (Participants) | 70 | 72 | 68
  Serotype 1:1 Month after Dose 4 | 162 [125 to 210] | 386 [306 to 486] | 194 [150 to 251]
  Serotype 3:1 Month after Dose 3: number analyzed (Participants) | 71 | 70 | 72
  Serotype 3:1 Month after Dose 3 | 107 [86 to 134] | 170 [147 to 196] | 120 [103 to 139]
  Serotype 3:Before Dose 4: number analyzed (Participants) | 70 | 70 | 69
  Serotype 3:Before Dose 4 | 16 [13 to 20] | 20 [16 to 25] | 16 [12 to 20]
  Serotype 3: 1 Month after Dose 4: number analyzed (Participants) | 68 | 70 | 66
  Serotype 3: 1 Month after Dose 4 | 131 [114 to 150] | 193 [165 to 226] | 150 [126 to 179]
  Serotype 4:1 Month after Dose 3: number analyzed (Participants) | 71 | 72 | 65
  Serotype 4:1 Month after Dose 3 | 1864 [1565 to 2219] | 1768 [1393 to 2245] | 1617 [1298 to 2015]
  Serotype 4: Before Dose 4: number analyzed (Participants) | 68 | 67 | 70
  Serotype 4: Before Dose 4 | 25 [18 to 37] | 44 [29 to 66] | 21 [15 to 28]
  Serotype 4:1 Month after Dose 4: number analyzed (Participants) | 70 | 71 | 67
  Serotype 4:1 Month after Dose 4 | 1627 [1232 to 2148] | 2038 [1471 to 2825] | 1544 [1224 to 1948]
  Serotype 5:1 Month after Dose 3: number analyzed (Participants) | 71 | 70 | 72
  Serotype 5:1 Month after Dose 3 | 95 [79 to 114] | 154 [131 to 183] | 91 [77 to 109]
  Serotype 5:Before Dose 4: number analyzed (Participants) | 71 | 71 | 71
  Serotype 5:Before Dose 4 | 16 [15 to 17] | 18 [16 to 19] | 15 [14 to 16]
  Serotype 5:1 Month after Dose 4: number analyzed (Participants) | 70 | 72 | 68
  Serotype 5:1 Month after Dose 4 | 172 [140 to 212] | 248 [204 to 303] | 141 [112 to 179]
  Serotype 6A:1 Month after Dose 3: number analyzed (Participants) | 71 | 70 | 72
  Serotype 6A:1 Month after Dose 3 | 2709 [2283 to 3213] | 3339 [2777 to 4013] | 3120 [2562 to 3799]
  Serotype 6A:Before Dose 4: number analyzed (Participants) | 67 | 70 | 66
  Serotype 6A:Before Dose 4 | 83 [56 to 122] | 173 [116 to 258] | 95 [62 to 147]
  Serotype 6A:1 Month after Dose 4: number analyzed (Participants) | 70 | 71 | 68
  Serotype 6A:1 Month after Dose 4 | 3249 [2686 to 3928] | 5455 [4379 to 6795] | 3489 [2831 to 4300]
  Serotype 6B:1 Month after Dose 3: number analyzed (Participants) | 70 | 69 | 72
  Serotype 6B:1 Month after Dose 3 | 1548 [1247 to 1921] | 2489 [2005 to 3088] | 1563 [1215 to 2010]
  Serotype 6B:Before Dose 4: number analyzed (Participants) | 68 | 65 | 70
  Serotype 6B:Before Dose 4 | 40 [29 to 54] | 75 [49 to 115] | 44 [31 to 63]
  Serotype 6B:1 Month after Dose 4: number analyzed (Participants) | 70 | 70 | 66
  Serotype 6B:1 Month after Dose 4 | 2304 [1811 to 2933] | 4319 [3478 to 5362] | 2552 [2006 to 3247]
  Serotype 7F:1 Month after Dose 3: number analyzed (Participants) | 69 | 74 | 69
  Serotype 7F:1 Month after Dose 3 | 4160 [3406 to 5081] | 4428 [3821 to 5131] | 4491 [3675 to 5490]
  Serotype 7F:Before Dose 4: number analyzed (Participants) | 65 | 70 | 69
  Serotype 7F:Before Dose 4 | 626 [436 to 899] | 761 [579 to 1000] | 689 [487 to 975]
  Serotype 7F:1 Month after Dose 4: number analyzed (Participants) | 70 | 71 | 67
  Serotype 7F:1 Month after Dose 4 | 4735 [3824 to 5863] | 6361 [5024 to 8054] | 4703 [3704 to 5972]
  Serotype 9V:1 Month after Dose 3: number analyzed (Participants) | 72 | 74 | 67
  Serotype 9V:1 Month after Dose 3 | 1807 [1432 to 2279] | 2388 [1986 to 2870] | 1929 [1554 to 2394]
  Serotype 9V:Before Dose 4: number analyzed (Participants) | 65 | 70 | 67
  Serotype 9V:Before Dose 4 | 183 [134 to 251] | 204 [151 to 274] | 212 [149 to 302]
  Serotype 9V:1 Month after Dose 4: number analyzed (Participants) | 70 | 70 | 68
  Serotype 9V:1 Month after Dose 4 | 4199 [3322 to 5309] | 5162 [4349 to 6127] | 4201 [3418 to 5164]
  Serotype 14:1 Month after Dose 3: number analyzed (Participants) | 70 | 69 | 72
  Serotype 14:1 Month after Dose 3 | 1922 [1429 to 2585] | 2593 [1999 to 3362] | 2103 [1527 to 2897]
  Serotype 14:Before Dose 4: number analyzed (Participants) | 68 | 71 | 68
  Serotype 14:Before Dose 4 | 426 [307 to 592] | 469 [346 to 634] | 357 [251 to 509]
  Serotype 14:1 Month after Dose 4: number analyzed (Participants) | 71 | 70 | 68
  Serotype 14:1 Month after Dose 4 | 1673 [1331 to 2102] | 1706 [1385 to 2102] | 2005 [1631 to 2463]
  Serotype 18C:1 Month after Dose 3: number analyzed (Participants) | 71 | 74 | 70
  Serotype 18C:1 Month after Dose 3 | 5124 [4381 to 5992] | 5355 [4617 to 6212] | 4908 [4037 to 5967]
  Serotype 18C:Before Dose 4: number analyzed (Participants) | 65 | 69 | 68
  Serotype 18C:Before Dose 4 | 122 [76 to 198] | 173 [112 to 267] | 89 [56 to 143]
  Serotype 18C:1 Month after Dose 4: number analyzed (Participants) | 70 | 70 | 66
  Serotype 18C:1 Month after Dose 4 | 4477 [3528 to 5681] | 6315 [5081 to 7848] | 4249 [3355 to 5381]
  Serotype 19A:1 Month after Dose 3: number analyzed (Participants) | 72 | 73 | 67
  Serotype 19A:1 Month after Dose 3 | 638 [535 to 762] | 676 [551 to 830] | 553 [441 to 693]
  Serotype 19A:Before Dose 4: number analyzed (Participants) | 67 | 71 | 67
  Serotype 19A:Before Dose 4 | 13 [10 to 18] | 20 [14 to 28] | 12 [10 to 16]
  Serotype 19A:1 Month after Dose 4: number analyzed (Participants) | 71 | 72 | 68
  Serotype 19A:1 Month after Dose 4 | 1860 [1530 to 2261] | 2534 [2044 to 3143] | 1722 [1379 to 2151]
  Serotype 19F:1 Month after Dose 3: number analyzed (Participants) | 71 | 70 | 71
  Serotype 19F:1 Month after Dose 3 | 449 [356 to 566] | 624 [494 to 788] | 488 [411 to 580]
  Serotype 19F:Before Dose 4: number analyzed (Participants) | 70 | 70 | 70
  Serotype 19F:Before Dose 4 | 26 [24 to 29] | 25 [24 to 26] | 26 [23 to 29]
  Serotype 19F:1 Month after Dose 4: number analyzed (Participants) | 71 | 71 | 68
  Serotype 19F:1 Month after Dose 4 | 1071 [846 to 1356] | 1783 [1364 to 2331] | 962 [753 to 1230]
  Serotype 23F:1 Month after Dose 3: number analyzed (Participants) | 72 | 74 | 71
  Serotype 23F:1 Month after Dose 3 | 1580 [1211 to 2061] | 1849 [1499 to 2281] | 1402 [1103 to 1782]
  Serotype 23F:Before Dose 4: number analyzed (Participants) | 64 | 70 | 66
  Serotype 23F:Before Dose 4 | 42 [24 to 73] | 62 [36 to 107] | 24 [15 to 39]
  Serotype 23F:1 Month after Dose 4: number analyzed (Participants) | 71 | 70 | 68
  Serotype 23F:1 Month after Dose 4 | 2609 [2015 to 3377] | 3772 [2966 to 4796] | 2052 [1668 to 2523]
  Serotype 8:1 Month after Dose 3: number analyzed (Participants) | 70 | 72 | 66
  Serotype 8:1 Month after Dose 3 | 1532 [1215 to 1933] | 16 [15 to 18] | 1541 [1220 to 1946]
  Serotype 8:Before Dose 4: number analyzed (Participants) | 65 | 73 | 65
  Serotype 8:Before Dose 4 | 166 [119 to 230] | 20 [17 to 24] | 147 [105 to 205]
  Serotype 8:1 Month after Dose 4: number analyzed (Participants) | 64 | 71 | 64
  Serotype 8:1 Month after Dose 4 | 2970 [2412 to 3658] | 27 [20 to 36] | 3208 [2525 to 4077]
  Serotype 10A:1 Month after Dose 3: number analyzed (Participants) | 63 | 75 | 63
  Serotype 10A:1 Month after Dose 3 | 6977 [5204 to 9354] | 40 [33 to 47] | 6780 [5436 to 8456]
  Serotype 10A:Before Dose 4: number analyzed (Participants) | 61 | 70 | 62
  Serotype 10A:Before Dose 4 | 1985 [1422 to 2772] | 78 [51 to 118] | 2066 [1439 to 2967]
  Serotype 10A:1 Month after Dose 4: number analyzed (Participants) | 61 | 68 | 58
  Serotype 10A:1 Month after Dose 4 | 9030 [6855 to 11893] | 87 [56 to 136] | 8269 [6252 to 10937]
  Serotype 11A:1 Month after Dose 3: number analyzed (Participants) | 73 | 73 | 67
  Serotype 11A:1 Month after Dose 3 | 1894 [1540 to 2330] | 58 [47 to 71] | 1838 [1451 to 2327]
  Serotype 11A:Before Dose 4: number analyzed (Participants) | 70 | 70 | 64
  Serotype 11A:Before Dose 4 | 416 [258 to 670] | 95 [64 to 142] | 247 [150 to 405]
  Serotype 11A: 1 Month after Dose 4: number analyzed (Participants) | 70 | 69 | 65
  Serotype 11A: 1 Month after Dose 4 | 3958 [2973 to 5269] | 90 [62 to 132] | 4200 [3187 to 5534]
  Serotype 12F:1 Month after Dose 3: number analyzed (Participants) | 46 | 75 | 44
  Serotype 12F:1 Month after Dose 3 | 35278 [23575 to 52790] | 24 [24 to 25] | 21475 [14378 to 32074]
  Serotype 12F:Before Dose 4: number analyzed (Participants) | 58 | 69 | 64
  Serotype 12F:Before Dose 4 | 3984 [3017 to 5261] | 35 [26 to 47] | 4904 [3909 to 6153]
  Serotype 12F:1 Month after Dose 4: number analyzed (Participants) | 57 | 74 | 47
  Serotype 12F:1 Month after Dose 4 | 15611 [11336 to 21499] | 43 [31 to 60] | 18899 [14215 to 25125]
  Serotype 15B:1 Month after Dose 3: number analyzed (Participants) | 71 | 74 | 66
  Serotype 15B:1 Month after Dose 3 | 6981 [5726 to 8511] | 17 [15 to 20] | 5707 [4129 to 7889]
  Serotype 15B:Before Dose 4: number analyzed (Participants) | 64 | 73 | 65
  Serotype 15B:Before Dose 4 | 578 [345 to 969] | 26 [18 to 39] | 609 [331 to 1121]
  Serotype 15B:1 Month after Dose 4: number analyzed (Participants) | 65 | 71 | 61
  Serotype 15B:1 Month after Dose 4 | 7280 [5594 to 9475] | 32 [20 to 50] | 7770 [6448 to 9363]
  Serotype 22F:1 Month after Dose 3: number analyzed (Participants) | 62 | 75 | 61
  Serotype 22F:1 Month after Dose 3 | 21864 [16413 to 29125] | 10 [8 to 11] | 19276 [14969 to 24822]
  Serotype 22F:Before Dose 4: number analyzed (Participants) | 66 | 72 | 64
  Serotype 22F:Before Dose 4 | 2562 [1869 to 3512] | 16 [11 to 24] | 2014 [1477 to 2745]
  Serotype 22F:1 Month after Dose 4: number analyzed (Participants) | 58 | 74 | 52
  Serotype 22F:1 Month after Dose 4 | 28435 [19414 to 41649] | 18 [12 to 27] | 23480 [17229 to 31998]
  Serotype 33F:1 Month after Dose 3: number analyzed (Participants) | 57 | 71 | 59
  Serotype 33F:1 Month after Dose 3 | 20162 [13581 to 29930] | 177 [160 to 195] | 15931 [11550 to 21974]
  Serotype 33F:Before Dose 4: number analyzed (Participants) | 56 | 72 | 60
  Serotype 33F:Before Dose 4 | 5678 [4403 to 7321] | 539 [391 to 742] | 6835 [5080 to 9198]
  Serotype 33F:1 Month after Dose 4: number analyzed (Participants) | 63 | 71 | 55
  Serotype 33F:1 Month after Dose 4 | 18997 [13140 to 27463] | 658 [480 to 904] | 26963 [18722 to 38830]

17. Secondary Outcome: Percentage of Participants With Pre-defined Pneumococcal Serotype-specific IgG Concentrations at 1 Month After Dose 4
Description: Pneumococcal serotype-specific IgG concentrations were measured for 20vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F. The predefined levels, >=0.35 micrograms/mL for all serotypes except for serotypes 5 (>=0.23 micrograms/mL), 6B (>=0.10 micrograms/mL) and 19A (>=0.12 micrograms/mL).
Time Frame: 1 Month after Dose 4
Population: Dose 4 evaluable immunogenicity population included participants who were eligible randomized aged 2 to 6 months of age at first dose, received all 4 randomized doses with Dose 4 received within defined window 12 to 15 months of age, had at least 1 immunogenicity results within 27 to 56 days, inclusive, after Dose 4,and had no other major protocol deviations per clinician. Here, N=participants evaluable for this outcome measure and n=participants with valid results for specified serotype.
Measure: Number; unit: Percentage of participants
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 217 | 220 | 211
Percentage of participants
  Serotype 1 | 99.1 | 100.0 | 98.6
  Serotype 3 | 91.7 | 98.6 | 91.5
  Serotype 4 | 100.0 | 100.0 | 100.0
  Serotype 5 | 99.5 | 100.0 | 99.5
  Serotype 6A | 100.0 | 100.0 | 100.0
  Serotype 6B: number analyzed (Participants) | 216 | 220 | 211
  Serotype 6B | 100.0 | 100.0 | 100.0
  Serotype 7F | 99.5 | 100.0 | 100.0
  Serotype 9V | 99.5 | 100.0 | 100.0
  Serotype 14 | 99.1 | 99.5 | 100.0
  Serotype 18C | 99.5 | 100.0 | 100.0
  Serotype 19A: number analyzed (Participants) | 217 | 219 | 211
  Serotype 19A | 100.0 | 100.0 | 100.0
  Serotype 19F | 100.0 | 100.0 | 100.0
  Serotype 23F | 99.5 | 100.0 | 99.5
  Serotype 8: number analyzed (Participants) | 217 | 219 | 211
  Serotype 8 | 100.0 | 3.2 | 100.0
  Serotype 10A | 99.1 | 0.9 | 99.5
  Serotype 11A | 100.0 | 5.9 | 100.0
  Serotype 12F | 98.2 | 0.0 | 98.6
  Serotype 15B | 100.0 | 8.6 | 100.0
  Serotype 22F | 100.0 | 1.8 | 100.0
  Serotype 33F | 100.0 | 2.7 | 100.0

18. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Serotype-Specific IgG Concentrations From 1 Month After Dose 3 to Before Dose 4
Description: GMFR of pneumococcal 20vPnC serotypes included: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F. The GMFR from 1 month after Dose 3 to before Dose 4 was reported from participants in Dose 3 evaluable immunogenicity population.
Time Frame: 1 Month after Dose 3 to before Dose 4
Population: Dose 3 evaluable immunogenicity population was included. Here, "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure and "Number Analyzed"= participants with valid IgG concentration at both timepoints for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 218 | 219 | 212
Fold rise
  Serotype 1 | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.2]
  Serotype 3 | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]
  Serotype 4 | 0.3 [0.2 to 0.3] | 0.2 [0.2 to 0.3] | 0.3 [0.2 to 0.3]
  Serotype 5: number analyzed (Participants) | 218 | 219 | 211
  Serotype 5 | 0.3 [0.2 to 0.3] | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.3]
  Serotype 6A | 0.5 [0.4 to 0.6] | 0.4 [0.4 to 0.4] | 0.4 [0.3 to 0.4]
  Serotype 6B: number analyzed (Participants) | 216 | 217 | 212
  Serotype 6B | 0.8 [0.6 to 0.9] | 0.5 [0.4 to 0.6] | 0.7 [0.6 to 0.8]
  Serotype 7F | 0.5 [0.4 to 0.5] | 0.4 [0.4 to 0.5] | 0.5 [0.4 to 0.5]
  Serotype 9V | 0.3 [0.2 to 0.3] | 0.3 [0.2 to 0.3] | 0.3 [0.2 to 0.3]
  Serotype 14: number analyzed (Participants) | 217 | 219 | 212
  Serotype 14 | 0.7 [0.6 to 0.8] | 0.7 [0.6 to 0.8] | 0.7 [0.6 to 0.8]
  Serotype 18C | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.2]
  Serotype 19A | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]
  Serotype 19F | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2]
  Serotype 23F | 0.2 [0.2 to 0.3] | 0.3 [0.2 to 0.3] | 0.3 [0.2 to 0.3]
  Serotype 8: number analyzed (Participants) | 218 | 216 | 212
  Serotype 8 | 0.2 [0.1 to 0.2] | 1.4 [1.2 to 1.6] | 0.2 [0.1 to 0.2]
  Serotype 10A | 2.2 [1.9 to 2.6] | 0.8 [0.6 to 0.9] | 2.3 [1.9 to 2.7]
  Serotype 11A | 0.1 [0.1 to 0.2] | 0.8 [0.6 to 0.9] | 0.1 [0.1 to 0.2]
  Serotype 12F | 0.4 [0.3 to 0.5] | 1.0 [0.9 to 1.1] | 0.4 [0.3 to 0.4]
  Serotype 15B | 0.4 [0.4 to 0.5] | 0.6 [0.5 to 0.7] | 0.4 [0.3 to 0.4]
  Serotype 22F | 0.4 [0.3 to 0.4] | 0.6 [0.5 to 0.8] | 0.4 [0.3 to 0.4]
  Serotype 33F: number analyzed (Participants) | 216 | 219 | 211
  Serotype 33F | 1.1 [0.9 to 1.2] | 0.6 [0.5 to 0.7] | 1.0 [0.9 to 1.2]

19. Secondary Outcome: GMFR in Serotype-Specific IgG Concentrations From 1 Month After Dose 3 to 1 Month After Dose 4
Description: GMFR of pneumococcal 20vPnC serotypes included: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F. The GMFR from 1 month after Dose 3 to 1 month after Dose 4 was reported from participants in both the Dose 3 and Dose 4 evaluable immunogenicity population.
Time Frame: From 1 Month after Dose 3 to 1 Month after Dose 4
Population: Dose 3 and Dose 4 evaluable immunogenicity populations were included. Here, "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure and "Number Analyzed"= participants with valid IgG concentrations at both timepoints for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 218 | 219 | 212
Fold rise
  Serotype 1: number analyzed (Participants) | 216 | 219 | 209
  Serotype 1 | 2.0 [1.8 to 2.2] | 2.1 [1.9 to 2.3] | 2.4 [2.2 to 2.7]
  Serotype 3: number analyzed (Participants) | 216 | 219 | 209
  Serotype 3 | 0.7 [0.7 to 0.8] | 0.8 [0.7 to 0.9] | 1.0 [0.9 to 1.1]
  Serotype 4: number analyzed (Participants) | 216 | 219 | 209
  Serotype 4 | 3.9 [3.4 to 4.4] | 3.4 [3.0 to 3.8] | 4.3 [3.7 to 4.8]
  Serotype 5: number analyzed (Participants) | 216 | 219 | 209
  Serotype 5 | 2.9 [2.6 to 3.3] | 2.7 [2.4 to 3.0] | 3.0 [2.6 to 3.4]
  Serotype 6A: number analyzed (Participants) | 216 | 219 | 209
  Serotype 6A | 8.6 [7.5 to 9.8] | 7.3 [6.5 to 8.3] | 8.6 [7.6 to 9.8]
  Serotype 6B: number analyzed (Participants) | 215 | 219 | 209
  Serotype 6B | 17.1 [14.3 to 20.4] | 12.6 [10.8 to 14.7] | 19.5 [16.2 to 23.5]
  Serotype 7F: number analyzed (Participants) | 216 | 219 | 209
  Serotype 7F | 2.8 [2.6 to 3.1] | 3.0 [2.7 to 3.3] | 3.3 [2.9 to 3.6]
  Serotype 9V: number analyzed (Participants) | 216 | 219 | 209
  Serotype 9V | 3.1 [2.8 to 3.5] | 3.1 [2.8 to 3.5] | 3.8 [3.4 to 4.2]
  Serotype 14: number analyzed (Participants) | 215 | 219 | 209
  Serotype 14 | 2.9 [2.6 to 3.4] | 3.1 [2.7 to 3.6] | 3.9 [3.3 to 4.5]
  Serotype 18C: number analyzed (Participants) | 216 | 219 | 209
  Serotype 18C | 2.3 [2.1 to 2.6] | 2.4 [2.1 to 2.6] | 2.5 [2.3 to 2.8]
  Serotype 19A: number analyzed (Participants) | 216 | 218 | 209
  Serotype 19A | 3.2 [2.8 to 3.6] | 2.8 [2.5 to 3.1] | 3.4 [3.0 to 3.8]
  Serotype 19F: number analyzed (Participants) | 216 | 219 | 209
  Serotype 19F | 3.1 [2.8 to 3.4] | 2.9 [2.6 to 3.3] | 3.1 [2.8 to 3.5]
  Serotype 23F: number analyzed (Participants) | 216 | 219 | 209
  Serotype 23F | 5.3 [4.6 to 6.1] | 5.7 [5.0 to 6.5] | 5.8 [5.1 to 6.6]
  Serotype 8: number analyzed (Participants) | 216 | 217 | 209
  Serotype 8 | 1.8 [1.6 to 2.0] | 1.7 [1.5 to 2.0] | 1.8 [1.6 to 2.0]
  Serotype 10A: number analyzed (Participants) | 216 | 219 | 209
  Serotype 10A | 14.0 [11.8 to 16.5] | 0.8 [0.7 to 1.0] | 17.5 [14.7 to 20.7]
  Serotype 11A: number analyzed (Participants) | 216 | 219 | 209
  Serotype 11A | 1.0 [0.9 to 1.1] | 0.8 [0.7 to 1.0] | 1.1 [1.0 to 1.2]
  Serotype 12F: number analyzed (Participants) | 216 | 219 | 209
  Serotype 12F | 3.4 [3.0 to 3.9] | 1.0 [1.0 to 1.1] | 3.9 [3.4 to 4.4]
  Serotype 15B: number analyzed (Participants) | 216 | 219 | 209
  Serotype 15B | 2.7 [2.4 to 3.1] | 0.9 [0.7 to 1.1] | 3.3 [2.9 to 3.7]
  Serotype 22F: number analyzed (Participants) | 216 | 219 | 209
  Serotype 22F | 2.9 [2.6 to 3.1] | 0.7 [0.6 to 0.9] | 3.2 [2.9 to 3.6]
  Serotype 33F: number analyzed (Participants) | 214 | 219 | 208
  Serotype 33F | 6.0 [5.3 to 6.7] | 0.7 [0.6 to 0.9] | 7.1 [6.2 to 8.1]

20. Secondary Outcome: GMFR in Serotype-Specific IgG Concentrations From Before Dose 4 to 1 Month After Dose 4
Description: GMFR of pneumococcal 20vPnC serotypes included: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F. The GMFR from before Dose 4 to 1 month after Dose 4 was reported from participants in the Dose 4 evaluable immunogenicity population.
Time Frame: From before Dose 4 to 1 Month after Dose 4
Population: Dose 4 evaluable immunogenicity population was included. Here, "Overall Number of Participants Analyzed" =participants evaluable for this outcome measure and "Number Analyzed" =participants with valid IgG concentrations at both timepoints for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
Number analyzed (Participants) | 217 | 220 | 211
Fold rise
  Serotype 1 | 10.7 [9.6 to 11.9] | 12.1 [11.0 to 13.3] | 12.6 [11.3 to 14.0]
  Serotype 3 | 7.5 [6.6 to 8.4] | 7.9 [7.1 to 8.8] | 8.9 [8.0 to 10.0]
  Serotype 4 | 15.0 [13.2 to 17.1] | 14.3 [12.7 to 16.0] | 16.5 [14.8 to 18.5]
  Serotype 5: number analyzed (Participants) | 217 | 220 | 210
  Serotype 5 | 10.8 [9.8 to 12.0] | 11.8 [10.7 to 13.1] | 12.2 [11.0 to 13.6]
  Serotype 6A | 17.6 [15.7 to 19.6] | 18.4 [16.6 to 20.5] | 22.1 [19.8 to 24.7]
  Serotype 6B: number analyzed (Participants) | 215 | 218 | 211
  Serotype 6B | 22.3 [19.9 to 24.9] | 24.3 [21.9 to 27.0] | 26.9 [23.9 to 30.2]
  Serotype 7F | 6.0 [5.5 to 6.6] | 7.2 [6.5 to 8.0] | 6.8 [6.2 to 7.5]
  Serotype 9V | 11.8 [10.5 to 13.2] | 12.0 [10.8 to 13.3] | 13.9 [12.4 to 15.6]
  Serotype 14 | 4.3 [3.8 to 4.9] | 4.4 [3.9 to 5.0] | 5.7 [5.0 to 6.6]
  Serotype 18C | 11.7 [10.5 to 12.9] | 14.0 [12.7 to 15.4] | 12.7 [11.5 to 14.1]
  Serotype 19A: number analyzed (Participants) | 217 | 219 | 211
  Serotype 19A | 34.2 [30.0 to 38.9] | 37.6 [33.2 to 42.6] | 38.3 [33.4 to 44.0]
  Serotype 19F | 18.8 [16.6 to 21.4] | 21.4 [19.0 to 24.2] | 19.9 [17.6 to 22.4]
  Serotype 23F | 22.6 [20.1 to 25.5] | 22.6 [19.8 to 25.7] | 22.7 [20.1 to 25.7]
  Serotype 8: number analyzed (Participants) | 217 | 218 | 211
  Serotype 8 | 10.8 [9.6 to 12.1] | 1.3 [1.2 to 1.4] | 11.2 [9.9 to 12.7]
  Serotype 10A | 6.3 [5.6 to 7.1] | 1.1 [1.0 to 1.1] | 7.4 [6.6 to 8.3]
  Serotype 11A | 7.0 [6.2 to 7.9] | 1.1 [1.0 to 1.2] | 8.1 [7.2 to 9.1]
  Serotype 12F | 8.5 [7.6 to 9.4] | 1.0 [1.0 to 1.1] | 9.9 [8.9 to 10.9]
  Serotype 15B | 6.8 [6.0 to 7.7] | 1.5 [1.3 to 1.6] | 8.7 [7.6 to 10.0]
  Serotype 22F | 7.9 [7.1 to 8.8] | 1.2 [1.1 to 1.3] | 8.9 [8.1 to 9.9]
  Serotype 33F | 5.7 [5.1 to 6.3] | 1.2 [1.1 to 1.3] | 6.9 [6.2 to 7.8]

ADVERSE EVENTS:
Time Frame: LR and SE [systematic assessment (SA)] within 7 days after Dose 1, 2, 3, or 4; SAEs (non-SA): from Day 1 up to 1 month after Dose 4; other AEs (non-SA): from Dose 1 up to 1 month after Dose 3 and from Dose 4 up to 1 month after Dose 4
Description: Same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be classified as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a SAE and non-SAE during the study
Arm/Group | 20vPnC (SC) | 13vPnC (SC) | 20vPnC (IM)
All-Cause Mortality (participants affected / at risk) | 0/225 | 0/224 | 1/217
Serious Adverse Events (participants affected / at risk) | 14/225 | 9/224 | 16/217
Other Adverse Events (participants affected / at risk) | 222/225 | 223/224 | 211/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20vPnC (SC) (N=225) | 13vPnC (SC) (N=224) | 20vPnC (IM) (N=217)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Congenital mitral valve incompetence (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Milk allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Exanthema subitum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 4 (4) | 2 (2) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Tuberculid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Kawasaki's disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20vPnC (SC) (N=225) | 13vPnC (SC) (N=224) | 20vPnC (IM) (N=217)
Injection site erythema (REDNESS) (General disorders) | 217 (762) | 217 (784) | 130 (297)
Injection site pain (PAIN) (General disorders) | 84 (167) | 85 (166) | 65 (118)
Injection site swelling (SWELLING) (General disorders) | 206 (723) | 211 (729) | 119 (251)
Pyrexia (FEVER) (General disorders) | 136 (219) | 135 (219) | 110 (197)
Bronchitis (Infections and infestations) | 8 (10) | 8 (9) | 11 (11)
Nasopharyngitis (Infections and infestations) | 49 (72) | 64 (85) | 66 (96)
Upper respiratory tract infection (Infections and infestations) | 12 (22) | 8 (10) | 8 (14)
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 62 (99) | 68 (118) | 55 (94)
Hypersomnia (INCREASED SLEEP) (Nervous system disorders) | 147 (343) | 161 (410) | 154 (389)
Irritability (IRRITABILITY) (Psychiatric disorders) | 110 (291) | 119 (295) | 107 (282)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 18 (22) | 11 (14) | 15 (19)
Eczema infantile (Skin and subcutaneous tissue disorders) | 6 (6) | 16 (18) | 13 (14)
Eczema (Skin and subcutaneous tissue disorders) | 22 (25) | 19 (19) | 32 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT04530838/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT04530838/SAP_001.pdf